CLINICAL TRIAL: NCT07060378
Title: A Study of Contrast-enhanced EBUS in Lung Lesions and Intrathoracic Lymph Nodes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Vice-President of the hospital, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KS25026
Record Dates: First submitted 2025-06-22; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-05

CONDITIONS: Lung Lesions; Mediastinal and Hilar Lymph Node Enlargement
Keywords: CE-EBUS; Ultrasound Contrast Agent; Microbubbles

STUDY DESIGN:
Intervention Model Description: Contrast-Enhanced Endobronchial Ultrasound
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contrast-Enhanced Endobronchial Ultrasound (Experimental)
  Interventions: Device: Contrast-enhanced endobronchial ultrasound

INTERVENTIONS:
Device: Contrast-enhanced endobronchial ultrasound — Using CE-EBUS to observe pulmonary lesions and abnormal enlarged intrathoracic lymph nodes, the enhancement characteristics of benign and malignant lesions under CE-EBUS were extracted for both conditions.

SUMMARY:
Exploring the Clinical Application Value of Contrast Enhancement Features in CE-EBUS Images for the Diagnosis of Pulmonary Lesions and Intrapulmonary Lymph Nodes

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old；
* Enlargement of at least one intrathoracic LN (short diameter > 1 cm) or central parenchymal lung lesions adjacent to the airway detected on chest CT, or increased fluorodeoxyglucose uptake in at least one intrathoracic lymph node on PET / CT (standardized uptake value > 2.5)；
* CP-EBUS-TBNA is required to determine the diagnosis or staging, the patient agreed to undergo CE-EBUS, and there were no contraindications to EBUS-TBNA;
* Patients who have good compliance and sign informed consent.

Exclusion Criteria:

* Patients with known hypersensitivity to ultrasound contrast components;
* Patients with severe pulmonary hypertension (pulmonary artery pressure > 90 mmHg);
* Patients with angina pectoris, acute coronary syndrome, clinically unstable ischemic heart disease, heart failure, cardiac dysfunction, and cardiac disease with right-to-left shunting;
* Patients with uncontrolled essential hypertension and adults with respiratory distress syndrome;
* Pregnant or lactating women；
* Patients with contraindications to bronchoscopy；
* Patients with other conditions that, in the opinion of the investigator, make the patient unsuitable for the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of CE-EBUS in the differential diagnosis of benign and malignant intrathoracic lymphadenopathy | 6 month post-procedure
  Diagnostic accuracy is defined as the number of lesions correctly identified as malignant or benign divided by the total number of lesions using CE-EBUS interpretation criteria.
Diagnostic accuracy of CE-EBUS in the differential diagnosis of benign and malignant intrapulmonary lesions | 6 month post-procedure
  Diagnostic accuracy was defined as the number of lesions correctly identified as malignant or benign divided by the total number of lesions using the CE-EBUS interpretation criteria.

SECONDARY OUTCOMES:
Sensitivity, specificity, positive predictive value and negative predictive value of CE-EBUS in the differential diagnosis of benign and malignant intrathoracic lymphadenopathy | 6 months post-procedure
  Sensitivity is defined as the number of lesions correctly identified as malignant using the CE-EBUS interpretation criteria divided by the total number of malignant lesions.
  Specificity is defined as the number of lesions correctly identified as benign using the CE-EBUS interpretation criteria divided by the total number of benign lesions.
  Positive predictive value is the percentage of truly malignant lesions among all lesions identified as malignant using the CE-EBUS interpretive criteria.
  Negative predictive value is the percentage of truly benign lesions among all lesions identified as benign using CE-EBUS interpretive criteria.
Sensitivity, specificity, positive predictive value and negative predictive value of CE-EBUS in the differential diagnosis of benign and malignant intrapulmonary lesions | 6 months post-procedure
  Sensitivity is defined as the number of lesions correctly identified as malignant using the CE-EBUS interpretation criteria divided by the total number of malignant lesions.
  Specificity is defined as the number of lesions correctly identified as benign using the CE-EBUS interpretation criteria divided by the total number of benign lesions.
  Positive predictive value is the percentage of truly malignant lesions among all lesions identified as malignant using the CE-EBUS interpretive criteria.
  Negative predictive value is the percentage of truly benign lesions among all lesions identified as benign using CE-EBUS interpretive criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGrath S, Shen YJ, Aragaki M, Motooka Y, Koga T, Gregor A, Bernards N, Cherin E, Demore CEM, Yasufuku K, Matsuura N. Imaging Microbubbles With Contrast-Enhanced Endobronchial Ultrasound. Ultrasound Med Biol. 2024 Jan;50(1):28-38. doi: 10.1016/j.ultrasmedbio.2023.08.020. Epub 2023 Oct 7. PMID 37813701
- [Background] Suriano I, Frasca L, Longo F, Sarubbi A, Tacchi G, Crucitti P. Diagnostic Yield of CE-EBUS in Mediastinal and Hilar Lymphadenopathy: A Preliminary Study. J Clin Med. 2025 Apr 18;14(8):2800. doi: 10.3390/jcm14082800. PMID 40283633